CLINICAL TRIAL: NCT07325916
Title: Relationship Between Serum Apolipoprotein Levels and Weight Loss in Patients Undergoing Sleeve Gastrectomy for Morbid Obesity
Status: Active, not recruiting | Type: Observational
Sponsor: Yigit DUZKOYLU (Other Government)
Responsible Party: Sponsor-Investigator, Yigit DUZKOYLU, Associate Professor, Başakşehir Çam & Sakura City Hospital
Organization: Başakşehir Çam & Sakura City Hospital (Other Government)
Other Study IDs: 2024-KAEK-11 134
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Morbid Obesity Requiring Bariatric Surgery
Keywords: morbid obesity; serum apolipoproteins; apolipoprotein AI; apolipoprotein AII; apolipoprotein B100; apolipoprotein CII; apolipoprotein CIII; apolipoprotein D; apolipoprotein E; apolipoprotein E4; apolipoprotein H; apolipoprotein J; apolipoprotein M; sleeve gastrectomy; bariatric surgery
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood will be centrifuged and serum will be stored separately in eppendorf tubes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sleeve Gastrectomy Patients: Patients who meet inclusion criteria for the study undergoing sleeve gastrectomy
  Interventions: Procedure: Laparoscopic Sleeve Gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic Sleeve Gastrectomy — Laparoscopic Sleeve Gastrectomy

SUMMARY:
The study looks at whether a specific protein in the blood, called apolipoprotein, can predict how much weight a person might lose after sleeve gastrectomy, a surgery for people with severe obesity. We want to find a specific level of this protein that shows which patients are most likely to lose weight successfully after surgery. By identifying this level, we hope to guide doctors in deciding who should have the surgery and who might do better with non-surgical weight loss methods.

DETAILED DESCRIPTION:
The subject of our research is whether serum apolipoprotein levels can be a predictive value for weight loss in patients who will undergo sleeve gastrectomy due to morbid obesity. Our aim is to determine a cut-off value for patients who benefit most from bariatric surgery based on preoperative serum apolipoprotein levels. By including this value among the surgical indications, we plan to direct patients less likely to benefit from surgery to conservative approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75
* International Classification of Diseases (ICD) code E66 diagnosis (obesity)
* Patients who have given consent for sleeve gastrectomy
* Patients who are suitable for general anesthesia

Exclusion Criteria:

* Patients who did not give consent to be included in the study
* Patients who are scheduled for surgery other than sleeve gastrectomy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients applying to Başakşehir Çam Sakura City Hospital General Surgery Clinic for bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in body mass index at 8 months | 8 months after surgery

SECONDARY OUTCOMES:
Change in lipid profile at 8 months | 8 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Cam and Sakura City Hospital, Istanbul, Basaksehir, Turkey (Türkiye)